CLINICAL TRIAL: NCT06564376
Title: Individually Tailored MgSo4 Supplementation to Reduce Cardiac and Renal Complications in Pediatric Heart Surgery
Brief Title: Tailored MgSO4 Supplementation to Reduce Complications in Pediatric Heart Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, David Rosen, MD, Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: s42qwux9
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: AKI - Acute Kidney Injury; Arrythmia; Congenital Heart Disease
Keywords: Acute Kidney Injury; Arrhythmias; Congenital heart surgery; Cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury; Arrhythmias, Cardiac; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Total magnesium (Other): Magnesium dosing based on total Mg blood level
  Interventions: Diagnostic Test: total magnesium
- ionized Magnesium (Active Comparator): Magnesium dosing based upon ionized Mg level
  Interventions: Device: ionized magnesium

INTERVENTIONS:
Diagnostic Test: total magnesium — Treatment based on total Magnesium
  Arms: Total magnesium
Device: ionized magnesium — Treatment based on ionized magnesium
  Arms: ionized Magnesium

SUMMARY:
Lay Summary

This study tests two ways of measuring blood magnesium after heart surgery. Children who need heart surgery may have heart and kidney problems after surgery. The right amount of magnesium in blood reduces this risk. This study will test the best way to measure magnesium. This will let doctors choose the right dose of MgSO4. MgSO4 is a magnesium supplement. Taking MgSO4 after heart surgery helps children. For each child, it is best to personalize MgSO4 dose. This is based on the amount of magnesium in blood. This study will test two ways of personalizing MgSO4 dose.

In the blood, there are two kinds of magnesium. Usually, blood magnesium tests measure both forms together. This does not say anything about active magnesium. This study will measure the two forms separately. Then, MgSO4 will be given based on either the active or whole magnesium. Measuring active magnesium is good. Active magnesium levels change faster than total. That means active magnesium tests may better protect children. Also, active magnesium has more of an impact on heart and kidney function. Focusing on the active form will help these organs stay healthy.

To test how well the MgSO4 is working, heart and kidneys will be examined. After surgery, certain harmful heart rhythms can occur. The types and number of harmful rhythms will be studied. Kidney problems can also happen after heart surgery. Kidney health will be studied. To help understand how active magnesium works, further tests will be done. These tests will look for evidence of poor health in the cells that make up the heart, kidney, and blood.

DETAILED DESCRIPTION:
Hypothesis: Modulating patient Mg levels based on ionized Mg will have clinical and functional benefits over using total Mg, due to the increased sensitivity and specificity of the ionized form. The primary goal of this project is to experimentally test the benefit of maintaining ionized normomagnesemia after cardiac surgery in children with regard to renal function and arrhythmia incidence . A secondary goal is to develop a model for predicting AKI after cardiac surgery in children, using a machine learning approach to understand interrelationships between magnesium-dependent physiological processes (Figure 1B). Successful completion of this project will define the utility and positionality of ionized Mg as an actor in pediatric post-surgical AKI, and its synergy with established clinical and physiological outcomes.

Aim 1: Investigating use of ionized Mg for Mg repletion therapy

In this aim, patients will be randomized to one of two strategies for Mg repletion therapy, one utilizing ionized Mg, the other using total Mg. The effects of these two strategies on clinical and physiological outcomes will be measured, as will the durability of the different Mg repletion strategies in preventing or correcting hypomagnesemia. 96 participants will be enrolled in this study. Because arrhythmia risk and AKI risk are dramatically stratified by age, subjects will be age-matched into the following groups: 0-1 month, 2 months to 2 years, 3- 9 years, 9 years -18 years. Children will be randomly assigned to one of two Mg repletion strategies. Randomization will occur after consenting and reaffirmation that the child/family/guardian still continue to agree to participate in the study. For each age group there will be 24 sealed envelopes that identify which treatment strategy for magnesium repletion they will be assigned (Total or ionized). This envelope will be opened at SBAR prior to the induction of anesthesia. Magnesium levels will be drawn and sent as per standard protocol. All patients will have ionized magnesium levels obtained with every blood gas, but only those in the ionized group will the physicians see and treat the magnesium based upon that value. Patients with hypomagnesemia ( value less than or equal to 1.8 Mg/dl in the total Magnesium group will be given MgSO4 at a standard dose of 50 mg/kg over 1 hour beginning at the intraoperative stage and at every subsequent timepoint where an individual's lab values show hypomagnesemia (Table 1). Those patients in the ionized magnesium group will be dosed according to Table 1 beginning at the intraoperative stage and at every subsequent timepoint where an individual's lab values show hypomagnesemia (Table 1). Study participants will be blinded to treatment group. Researchers will not be blinded at the time of MgSO4 administration due to logistical pharmacy requirements. All data analysis including ECG analysis will be performed by blinded researchers. In one arm, Mg repletion will be titrated using ionized Mg as a measure, maintaining an ionized Mg level of 0.98-1.46 mg/dl. In the other, Mg repletion will be titrated using total Mg as a measure. Due to reagents used by WVU labs, the reference range for total Mg is 1.9-3.1 mg/dL; patients in the total Mg arm will be maintained in this range. To ensure proper electrolyte balance, Ca2+, K+, and Na+ will be maintained within appropriate ranges using standard methodology.

Mg level will be measured on all arterial blood gases. Mg will be measured at least: pre-incision, at the completion of the procedure, and twice a day for 48 hours after surgery. In order to assess differences in post-treatment Mg maintenance after cessation of therapy, ionized and total Mg levels will also be measured 4 hours after Mg supplementation.

Urinary NGAL and Creatinine will be measured pre-bypass, 2 hours after bypass and 24 hours after bypass to assess for renal injury.

Clinical outcomes to be measured include:

1. Urine output, measured hourly for 48 hours after surgery.
2. Blood lactate, measured at least daily (standard of care).
3. Time to extubation.
4. Occurrence of non-sinus cardiac rhythms, with special attention given to accelerated junctional rhythms.

Magnesium dosing Total Mg (mg/dL) Less than or equal to 1.8 MgSO4 dose 50 mg/kg Ionized Mg Observed Mg(Mg/dL) MgSO4 dose 1.3 10 mg/kg - 1 hr 1.2 20 mg/kg - 1 hr 1.0 30 mg/kg - 1 hr 0.9 40 mg/kg - 1 hr 0.8 50 mg/kg - 1hr

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing cardiac surgery utilizing cardiopulmonary bypass

Exclusion Criteria:

* Children undergoing cardiac surgery without cardiopulmonary bypass
* Children with Renal disease
* Children with pre-existing arrhythmia
* Children on anti-arrhythmia medication

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Duration from reanimation to sinus rhythm | 48 hours after reanimation
Time in non-sinus rhythms: within 24h of removing aortic cross-clamp | first 24 hours after reanimation
Time in non-sinus rhythms: 24-48h after removing aortic cross-clamp | 24-48 hours after reanimation
Presence of any arrhythmia | 48 hours after reanimation
  Defined as any non-sinus rhythm
Urine NGAL concentration | 48 hours after reanimation
  Sensitive marker of acute kidney injury
Urine Creatinine concentration | 48 hours after reanimation
  The combination of NGAL/Creatine increases sensitivity marker of acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: David A Rosen, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States